CLINICAL TRIAL: NCT03441984
Title: A 2-Part, Phase I, Single-Dose, 3-Period Crossover Relative Bioavailability Study of a Pediatric TRIUMEQ Dispersible Tablet and Pediatric Dolutegravir and Lamivudine (DTG/3TC) Fixed Dose Combination Dispersible Tablet Formulations as Compared With Adult Tablets in Healthy Volunteers
Brief Title: To Assess the Relative Bioavailability (BA) of TRIUMEQ® and Dolutegravir and Lamivudine (DTG/3TC) Pediatric Dispersible Tablet Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry); Pharmaceutical Product Development (PPD), Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205894
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: HIV Infections
Keywords: Pediatric dispersible tablets; Bioavailability
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: 2-part study with 3-TPs each. Part 1, compares relative BA of TRIUMEQ dispersible tablets for pediatric populations (DTG, 5 milligram [mg]/abacavir [ABC] 60 mg/3TC 30 mg), when administered as direct-to-mouth and when dispersed into purified water, with adult TRIUMEQ conventional tablet (DTG 50 mg/ABC 600 mg/3TC 300 mg), administered as direct-to-mouth (reference). Additionally, part 2 will compare relative BA of DTG/3TC (DTG 5 mg/3TC 30 mg), dispersible tablets for pediatric populations, when administered as direct-to mouth and when dispersed into purified water, with adult DTG (50 mg) and 3TC (300 mg) conventional tablets, when administered as direct-to-mouth (reference). Each TP, in Part 1 and 2 will have, wash-out period of 7-days (with minus 4 hours) between each single dose, for flexible dosing. During TPs, subjects will be admitted, to clinic on Day-1, following completion of last study procedure on Day 4, post which follow-up visit conducted, 7 to 10 days after last dose.
Masking Description: This is an open-label study in healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Subjects with treatment sequence ABC (Experimental): The subjects in Part 1 of the study, will receive a single dose of treatment A= adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, 1 conventional tablet) administered as direct-to-mouth, in TP1; treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately in TP2; and treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence BCA (Experimental): The subjects in Part 1 of the study, will receive treatment B in TP1, treatment C in TP2 and treatment A in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence CAB (Experimental): The subjects in Part 1 of the study will receive a single dose each of, treatment C in TP1, treatment A in TP2 and treatment B in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence ACB (Experimental): The subjects in Part 1 of the study will receive, treatment A in TP1, treatment C in TP2 and treatment B in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence BAC (Experimental): The subjects in Part 1 of the study will receive a single dose each of, treatment B in TP1, treatment A in TP2 and treatment C in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence CBA (Experimental): The subjects in Part 1 of the study will receive a single dose each of, treatment C in TP1, treatment B in TP2 and treatment A in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Subjects with treatment sequence DEF (Experimental): The subjects in Part 2 of the study, will receive a single dose of treatment D= Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg, 1 conventional tablet) administered as direct-to-mouth, in TP1; treatment E= Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately in TP2; and treatment F= Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Subjects with treatment sequence EFD (Experimental): The subjects in Part 2 of the study, will receive a single dose respectively of treatment E in TP1, treatment F in TP2 and treatment D in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Subjects with treatment sequence FDE (Experimental): The subjects in Part 2 of the study, will receive a single dose of treatment F in TP1, treatment D in TP2 and treatment E in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Subjects with treatment sequence DFE (Experimental): The subjects in Part 2 of the study, will receive a single dose of treatment D in TP1, treatment F in TP2 and treatment E in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Subjects with treatment sequence EDF (Experimental): The subjects in Part 2 of the study, will receive a single dose of treatment E in TP1, treatment D in TP2 and treatment F in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Subjects with treatment sequence FED (Experimental): The subjects in Part 2 of the study, will receive a single dose of treatment F in TP1, treatment E in TP2 and treatment D in TP3. Each treatment will be followed by a wash-out period of 7-days minus 4 hours.
  Interventions: Drug: Treatment D; Drug: Treatment F

INTERVENTIONS:
Drug: Treatment A — TRIUMEQ (Adult) administered as a, single dose, fixed dose combination (FDC) tablet - DTG 50 mg/ABC 600 mg/3TC 300 mg as 1 conventional tablet, orally as direct-to-mouth.
  Arms: Subjects with treatment sequence ABC; Subjects with treatment sequence ACB; Subjects with treatment sequence BAC; Subjects with treatment sequence BCA; Subjects with treatment sequence CAB; Subjects with treatment sequence CBA
Drug: Treatment B — TRIUMEQ (Pediatric) administered as a, single dose, FDC tablet - DTG 5 mg/ABC 60 mg/ 3TC 30 mg, orally as 10 dispersible tablets
  Arms: Subjects with treatment sequence ABC; Subjects with treatment sequence ACB; Subjects with treatment sequence BAC; Subjects with treatment sequence BCA; Subjects with treatment sequence CAB; Subjects with treatment sequence CBA
Drug: Treatment C — TRIUMEQ (Pediatric) administered as a, single dose, FDC tablet - DTG 5 mg/ABC 60 mg/3TC 30 mg, orally as direct-to-mouth.
  Arms: Subjects with treatment sequence ABC; Subjects with treatment sequence ACB; Subjects with treatment sequence BAC; Subjects with treatment sequence BCA; Subjects with treatment sequence CAB; Subjects with treatment sequence CBA
Drug: Treatment D — DTG and 3TC (Adult), administered as a, single dose, Single dose, 1 tablet DTG (50 mg) and
  1 tablet 3TC (300 mg), orally as direct-to-mouth.
  Arms: Subjects with treatment sequence DEF; Subjects with treatment sequence DFE; Subjects with treatment sequence EDF; Subjects with treatment sequence EFD; Subjects with treatment sequence FDE; Subjects with treatment sequence FED
Drug: Treatment E — DTG and 3TC (Pediatric) administered as a, single dose, FDC tablet single dose, FDC tablet - DTG 5 mg/3TC 30 mg, orally as 10 dispersible tablets.
  Arms: Subjects with treatment sequence DEF; Subjects with treatment sequence DFE; Subjects with treatment sequence EDF; Subjects with treatment sequence EFD; Subjects with treatment sequence FDE
Drug: Treatment F — DTG and 3TC (Pediatric) administered as a, single dose, FDC tablet single dose, FDC tablet - DTG 5 mg/3TC 30 mg, orally as direct-to-mouth.
  Arms: Subjects with treatment sequence DEF; Subjects with treatment sequence DFE; Subjects with treatment sequence EDF; Subjects with treatment sequence EFD; Subjects with treatment sequence FDE; Subjects with treatment sequence FED

SUMMARY:
This is a 2-part, single-dose, open label, randomized 3-way cross-over study to compare BA of pediatric study drugs TRIUMEQ and (DTG/3TC) in healthy volunteers under fasted conditions. Study will be conducted in 2-parts. Each part 1 and part 2 will comprise of 3-treatment periods (TP) where Part 1, will assess BA, of pediatric TRIUMEQ dispersible tablets with an adult TRIUMEQ conventional tablet formulation and Part 2, will assess BA, of pediatric DTG/3TC dispersible tablets with adult DTG and 3TC conventional tablets formulation. Total duration of study is 9-weeks and will be conducted in approximately 36 subjects. The 2-parts, may be run in parallel as they are independent of each other. TRIUMEQ is a registered trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age, inclusive, at the time of signing the informed consent.
* Healthy subjects as determined by the investigator or medically qualified designee based on a medical evaluation, including medical history, physical examination, laboratory tests, and cardiac evaluation (history and ECG).
* Body weight >=50 kilogram (kg) for males and >=45 kg for females and body mass index (BMI) within the range 18.5 - 31.0 kilogram per square meter (kg/m^2) (inclusive).
* Male and female subjects where the male subjects must agree to use contraception during the TP and for at least 2 weeks plus an additional 90 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period. For the female subjects, female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least 1 of the following conditions applies: Female with non-reproductive potential, defined as Premenopausal females with one of the following like documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, documented hysterectomy, documented bilateral oophorectomy, the Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT), and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment; Females with reproductive potential and agrees to follow one of the options for avoiding pregnancy in females of reproductive potential, from 30 days prior to the first dose of study medication and until 2 weeks after dosing with study medication and completion of the follow-up visit; the investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception; All female subjects participating in the study should be counselled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of human immune virus (HIV) transmission to an uninfected partner.
* Subjects capable of giving signed informed consent.
* For participation in Part 1, documentation that the subject is negative for the human leukocyte antigen (HLA)-B*5701 allele.

Exclusion Criteria:

* The medical conditions included where ALT and bilirubin >1.5 × upper limit of normal (ULN) (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < =35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) where the heart rate for the male subjects be <45 and >100 beats per minute (bpm) and that for females be < 50 and > 100 bpm; the PR interval for both be < 120 and > 220 millisecond (msec); the QRS interval be < 70 and > 120 msec and the corrected Q-T interval (QTc) obtained using the Fridericia's formula (QTcF) be >450 msec ; ECG with evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization; any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [2nd degree or higher], Wolf-Parkinson-White syndrome); Sinus pauses > 3 seconds; any significant arrhythmia which, in the opinion of the principal investigator or ViiV/GlaxoSmithKline (GSK) medical monitor, will interfere with the safety of the individual subject; non-sustained or sustained ventricular tachycardia (3 consecutive ventricular ectopic beats).
* Subjects with use of prior or concomitant therapy who are unable to refrain from the use of prescription (e.g., dofetilide) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and ViiV Healthcare Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >14 drinks for males or > 7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine, or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 1 month prior to screening.
* Contraindications like history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation. The subject has participated in a clinical trial and has received an investigational product (IP) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the IP (whichever is longer).
* The subject has participated in a clinical trial and has received an IP within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the IP (whichever is longer).
* Creatinine clearance (CrCL) < 90 mL per minute.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol/cotinine screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 60 days.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has submitted approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Singh RP, Adkison KK, Baker M, Parasrampuria R, Wolstenholme A, Davies M, Sewell N, Brothers C, Buchanan AM. Development of Dolutegravir Single-entity and Fixed-dose Combination Formulations for Children. Pediatr Infect Dis J. 2022 Mar 1;41(3):230-237. doi: 10.1097/INF.0000000000003366. PMID 34817414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-Part, Phase I, Single-Dose, 3-Period Crossover Relative Bioavailability Study of a Pediatric TRIUMEQ Dispersible Tablet and Pediatric Dolutegravir and Lamivudine (DTG/3TC) Fixed Dose Combination Dispersible Tablet Formulations as Compared with Adult Tablets in Healthy Participants.
Pre-assignment Details: A total of 36 participants were enrolled for Part 1 and 2 of the study at a single-center in the United States. Each participant received all 3 treatments according to their assignment to one of the 6 treatment sequences in Part 1 and 2.
Groups:
- Treatment Sequence ABC-Part 1: Participants received either treatment A=Adult TRIUMEQ (Dolutegravir [DTG] 50 milligram [mg]/Abacavir [ABC] 600 mg/Lamivudine [3TC] 300 mg, one tablet) direct-to-mouth or treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion or treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth followed by a wash-out period of 7 days after each treatment.
- Treatment Sequence BCA-Part 1: Participants received either treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion or treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth or treatment A=Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, one tablet) direct-to-mouth followed by a wash-out period of 7 days.
- Treatment Sequence CAB-Part 1: Participants received either treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth or treatment A=Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, one tablet) direct-to-mouth or treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion followed by a wash-out period of 7 days.
- Treatment Sequence ACB-Part 1: Participants received either treatment A=Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, one tablet) direct-to-mouth or treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth or treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion followed by a wash-out period of 7 days.
- Treatment Sequence BAC-Part 1: Participants received either treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion or treatment A=Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, one tablet) direct-to-mouth or treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth followed by a wash-out period of 7 days.
- Treatment Sequence CBA-Part 1: Participants received either treatment C=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) direct-to-mouth or treatment B=Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) as a dispersion or treatment A=Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg. one tablet) direct-to-mouth followed by a wash-out period of 7 days.
- Treatment DEF-Part 2: Participants received either treatment D=Adult DTG 50 mg and 3TC 300 mg as one conventional tablet direct-to-mouth or treatment E=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets as dispersion or treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth followed by a wash-out period of 7 days.
- Treatment EFD-Part 2: Participants received either treatment E=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets as dispersion or treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth or treatment D=Adult DTG 50 mg and 3TC 300 mg as one conventional tablet direct-to-mouth followed by a wash-out period of 7 days.
- Treatment FDE-Part 2: Participants received either treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth or treatment D=Adult DTG 50 mg and 3TC 300 mg, one conventional tablet direct-to-mouth or treatment E=Pediatric DTG 5 mg/3TC 30 mg, as 10 dispersible tablets as dispersion followed by a wash-out period of 7 days.
- Treatment DFE-Part 2: Participants received either treatment D=Adult DTG 50 mg and 3TC 300 mg, as one conventional tablet direct-to-mouth or treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth or treatment E=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets as dispersion followed by a wash-out period of 7 days.
- Treatment EDF-Part 2: Participants received either treatment E=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets as dispersion or treatment D=Adult DTG 50 mg and 3TC 300 mg, one coventional tablet direct-to-mouth or treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth followed by a wash-out period of 7 days.
- Treatment FED-Part 2: Participants received either treatment F=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets direct-to-mouth or treatment E=Pediatric DTG 5 mg/3TC 30 mg, 10 dispersible tablets as dispersion or treatment D=Adult DTG 50 mg and 3TC 300 mg, one conventional tablet direct-to-mouth followed by a wash-out period of 7 days.
Period: Part 1: Period 1 (Up to Day 4)
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1,Period 1: Wash-out Period: 7 Days
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2 (Up to Day 4 )
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Positive urine drug screen lab value | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2,Wash-out Period: 7 Days
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 3 (Up to Day 4 )
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 1(Up to Day 4)
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 1, Wash-out: Up to 7 Days
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 2 (Up to Day 4)
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 2, Wash-out: Up to 7 Days
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 3 (Up to Day 4)
Arm/Group | Treatment Sequence ABC-Part 1 | Treatment Sequence BCA-Part 1 | Treatment Sequence CAB-Part 1 | Treatment Sequence ACB-Part 1 | Treatment Sequence BAC-Part 1 | Treatment Sequence CBA-Part 1 | Treatment DEF-Part 2 | Treatment EFD-Part 2 | Treatment FDE-Part 2 | Treatment DFE-Part 2 | Treatment EDF-Part 2 | Treatment FED-Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants in Part 1: All participants received either treatment A or B or C in 6 treatment sequences: ABC, BCA, CAB, ACB, CBA and BAC
- All Study Participants in Part 2: All participants received either treatment D or E or F in 6 treatment sequences: DEF, EFD, FDE, DFE, EDF and FED
- Total: Total of all reporting groups
Arm/Group | All Study Participants in Part 1 | All Study Participants in Part 2 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (10.08) | 33.9 (8.47) | 34.4 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian-Central/South Asian Heritage | 0 | 0 | 0
  Asian-Japanese/East/South-East Asian Heritage | 0 | 4 | 4
  Black or African American | 5 | 6 | 11
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time of Dose Extrapolated to Infinity (AUC[0-inf]) in Part 1 of DTG
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate pharmacokinetic (PK) parameters of DTG in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods. PK population comprised of participants in the all participants population (participants who took at least 1 dose of study medication) for whom PK sample was obtained and who had evaluable PK assay results. Statistics has been presented on geometric least square (LS) means.
Time Frame: Pre-dose, 15 and 30 minutes, 1 , 1.5 , 2 , 2.5 , 3 , 4 , 5 , 6 , 8 , 12 , 16 , 24 , 48 and 72 hours post-dose of each treatment period
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet: Participants received adult TRIUMEQ as 1 conventional tablet administered as direct-to-mouth.
- DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets: Participants received pediatric TRIUMEQ as 10 dispersible tablets administered as dispersion and taken immediately.
- DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth: Participants received pediatric TRIUMEQ as 10 dispersible tablets administered as direct-to-mouth.
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 59.761 (31) | 101.125 (22) | 77.742 (29)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.6946, 90% CI 2-sided [1.5690 to 1.8373] — Treatment comparison of pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg dispersible tablets) and adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg tablet) is presented
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.3512, 90% CI 2-sided [1.2465 to 1.4647] — Treatment comparison of pediatric TRUMEQ (DTG 5 mg/ABC 60 mg/3TC 30mg dispersible tablet direct to mouth) and adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg tablet) is presented
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2541, 90% CI 2-sided [1.1569 to 1.3595] — Treatment comparison of pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg dispersible tablets) and pediatric TRUMEQ (DTG 5 mg/ABC 60 mg/3TC 30mg dispersible tablet direct to mouth) is presented

2. Primary Outcome: AUC From Time of Dose to Last Measurable Concentration (AUC[0-t]) in Part 1 of DTG
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: Pre-dose,15 and 30 minutes,1 ,1.5 ,2 ,2.5 ,3 ,4 ,5 ,6 ,8 ,12 ,16 ,24 ,48 and 72 hours post-dose of each treatment period
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 57.571 (29) | 97.746 (21) | 75.086 (28)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.7001, 90% CI 2-sided [1.5685 to 1.8428] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.3519, 90% CI 2-sided [1.2475 to 1.4650] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2576, 90% CI 2-sided [1.1605 to 1.3629] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Maximum Observed Concentration (Cmax) in Part 1 of DTG in Plasma
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 1. PK analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Micrograms per milliliter | 3.093 (20) | 5.373 (15) | 4.134 (21)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.7382, 90% CI 2-sided [1.5983 to 1.8904] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.3614, 90% CI 2-sided [1.2525 to 1.4798] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2768, 90% CI 2-sided [1.1746 to 1.3878] — [estimate comment as in outcome 1, analysis 3]

4. Primary Outcome: AUC(0-inf) in Part 1 of ABC
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of ABC in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 16.636 (21) | 17.321 (20) | 16.756 (22)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0407, 90% CI 2-sided [1.0118 to 1.0704] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0228, 90% CI 2-sided [0.9944 to 1.0520] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0175, 90% CI 2-sided [0.9893 to 1.0465] — [estimate comment as in outcome 1, analysis 3]

5. Primary Outcome: AUC(0-t) in Part 1 of ABC
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of ABC in Part 1. PK analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 16.609 (21) | 17.298 (20) | 16.735 (22)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0410, 90% CI 2-sided [1.0121 to 1.0708] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0232, 90% CI 2-sided [0.9948 to 1.0524] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0174, 90% CI 2-sided [0.9892 to 1.0465] — [estimate comment as in outcome 1, analysis 3]

6. Primary Outcome: Cmax in Part 1 of ABC in Plasma
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Micrograms per milliliter | 5.084 (19) | 5.351 (19) | 4.891 (23)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0533, 90% CI 2-sided [0.9885 to 1.1223] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9766, 90% CI 2-sided [0.9167 to 1.0405] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0785, 90% CI 2-sided [1.0123 to 1.1490] — [estimate comment as in outcome 1, analysis 3]

7. Primary Outcome: AUC(0-inf) in Part 1 of 3TC
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of 3TC in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 13.087 (26) | 13.062 (24) | 12.155 (30)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0000, 90% CI 2-sided [0.9536 to 1.0486] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9478, 90% CI 2-sided [0.9039 to 0.9939] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0550, 90% CI 2-sided [1.0061 to 1.1063] — [estimate comment as in outcome 1, analysis 3]

8. Primary Outcome: AUC (0-t) in Part 1 of 3TC
Description: as for outcome 7
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 12.857 (26) | 12.829 (24) | 11.893 (29)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 0.9994, 90% CI 2-sided [0.9525 to 1.0486] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9432, 90% CI 2-sided [0.8990 to 0.9896] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0596, 90% CI 2-sided [1.0099 to 1.1117] — [estimate comment as in outcome 1, analysis 3]

9. Primary Outcome: Cmax in Part 1 of 3TC
Description: as for outcome 7
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Micrograms per milliliter | 2.194 (29) | 2.053 (35) | 1.947 (34)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 0.9362, 90% CI 2-sided [0.8677 to 1.0101] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9079, 90% CI 2-sided [0.8416 to 0.9795] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0312, 90% CI 2-sided [0.9558 to 1.1124] — [estimate comment as in outcome 1, analysis 3]

10. Primary Outcome: AUC(0-inf) in Part 2 of DTG in Plasma
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 2. PK analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- DTG 50 mg/3TC 300 mg Tablet: Participants received adult DTG and 3TC as one conventional tablet direct-to-mouth
- DTG 5 mg/3TC 30 mg Dispersible Tablet: Participants received 10 dispersible pediatric DTG/3TC tablets as dispersion
- DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth: Participants received 10 dispersible pediatric DTG/3TC tablets direct-to-mouth
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 53.942 (38) | 88.676 (31) | 68.496 (32)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 1.6439, 90% CI 2-sided [1.4649 to 1.8449] — Treatment comparison of pediatric DTG/3TC (DTG 5 mg/3TC 30 mg dispersible tablet) and adult DTG/3TC (DTG 50 mg/3TC 300 mg tablet) is presented
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2698, 90% CI 2-sided [1.1315 to 1.4250] — Treatment comparison of pediatric DTG/3TC (DTG 5 mg/3TC 30 mg dispersible tablet direct to mouth) and pediatric DTG/3TC (DTG 5 mg/3TC 30 mg dispersible tablet) is presented
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2946, 90% CI 2-sided [1.1536 to 1.4529] — Treatment comparison of pediatric DTG/3TC (DTG 5 mg/3TC 30 mg dispersible tablet direct to mouth) and pediatric DTG/3TC (DTG 5 mg/3TC 30 mg dispersible tablet direct to mouth) is presented

11. Primary Outcome: AUC(0-t) in Part 2 of DTG
Description: as for outcome 10
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 51.477 (38) | 85.340 (30) | 65.657 (31)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 1.6578, 90% CI 2-sided [1.4709 to 1.8685] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2755, 90% CI 2-sided [1.1317 to 1.4375] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2998, 90% CI 2-sided [1.1533 to 1.4650] — [estimate comment as in outcome 10, analysis 3]

12. Primary Outcome: Cmax in Part 2 of DTG in Plasma
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Micrograms per milliliter | 2.764 (44) | 5.461 (18) | 3.558 (28)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 1.9758, 90% CI 2-sided [1.7585 to 2.2201] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2873, 90% CI 2-sided [1.1457 to 1.4465] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.5348, 90% CI 2-sided [1.3660 to 1.7245] — [estimate comment as in outcome 10, analysis 3]

13. Primary Outcome: AUC(0-inf) in Part 2 of 3TC
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of 3TC in Part 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 12.245 (17) | 12.149 (21) | 11.910 (20)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 0.9798, 90% CI 2-sided [0.9241 to 1.0389] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9605, 90% CI 2-sided [0.9059 to 1.0185] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0201, 90% CI 2-sided [0.9633 to 1.0802] — [estimate comment as in outcome 10, analysis 3]

14. Primary Outcome: AUC(0-t) in Part 2 of 3TC
Description: as for outcome 13
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 11.991 (16) | 11.788 (20) | 11.633 (19)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 0.9831, 90% CI 2-sided [0.9243 to 1.0457] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9702, 90% CI 2-sided [0.9121 to 1.0320] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0134, 90% CI 2-sided [0.9527 to 1.0779] — [estimate comment as in outcome 10, analysis 3]

15. Primary Outcome: Cmax in Part 2 of 3TC
Description: as for outcome 7
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Micrograms per milliliter | 2.276 (28) | 2.071 (27) | 2.093 (29)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 0.9100, 90% CI 2-sided [0.8196 to 1.0102] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9198, 90% CI 2-sided [0.8285 to 1.0212] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9893, 90% CI 2-sided [0.8911 to 1.0983] — [estimate comment as in outcome 10, analysis 3]

16. Secondary Outcome: AUC From Time of Dose to 24 Hours (AUC[0-24]) of DTG in Part 1
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 15 and 30 minutes, 1 , 1.5 , 2 , 2.5 , 3 , 4 , 5 , 6 , 8 , 12 , 16 and 24 hours post-dose of each treatment period
Population: PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 40.264 (23) | 69.745 (17) | 53.250 (22)

17. Secondary Outcome: Time to Maximum Concentration (Tmax) of DTG in Plasma in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 3.00 [1.50 to 4.08] | 2.50 [1.00 to 6.00] | 3.00 [1.00 to 6.00]

18. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast) of DTG in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population.
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 72.00 [72.00 to 72.00] | 72.00 [72.00 to 72.30] | 72.00 [72.00 to 72.02]

19. Secondary Outcome: Apparent Oral Clearance (CL/F) of DTG in Plasma in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters per hour | 0.8367 (31) | 0.4944 (22) | 0.6432 (29)

20. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of DTG in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters | 17.260 (20) | 10.074 (20) | 12.998 (21)

21. Secondary Outcome: Observed Concentration at 24 Hours Postdose (C24) of DTG in Plasma in Part 1
Description: as for outcome 2
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per millilter | 925.303 (34) | 1523.534 (28) | 1198.948 (33)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.6503, 90% CI 2-sided [1.5131 to 1.8000] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.3501, 90% CI 2-sided [1.2381 to 1.4722] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2224, 90% CI 2-sided [1.1210 to 1.3330] — [estimate comment as in outcome 1, analysis 3]

22. Secondary Outcome: Last Observed Quantifiable Concentration (Ct) of DTG in Plasma in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per milliliter | 84.968 (83) | 138.258 (65) | 106.140 (80)

23. Secondary Outcome: Terminal Elimination Phase Half-life (t½) of DTG in Plasma in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 14.300 (21) | 14.123 (18) | 14.008 (20)

24. Secondary Outcome: Lag Time for Absorption (Tlag) of DTG in Part 1
Description: as for outcome 16
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 0.00 [0.00 to 0.25] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

25. Secondary Outcome: AUC(0-24) of ABC in Plasma in Part 1
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of ABC in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 16.619 (21) | 17.300 (20) | 16.743 (22)

26. Secondary Outcome: Tmax of ABC in Plasma in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 1.50 [0.50 to 2.57] | 1.00 [0.25 to 2.00] | 1.00 [0.25 to 2.00]

27. Secondary Outcome: Tlast of ABC in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 24.00 [16.00 to 24.07] | 24.00 [16.00 to 24.12] | 24.00 [16.00 to 24.07]

28. Secondary Outcome: CL/F of ABC in Plasma in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters per hour | 36.0658 (21) | 34.6391 (20) | 35.8073 (22)

29. Secondary Outcome: Vz/F of ABC in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters | 120.412 (46) | 126.171 (39) | 123.076 (42)

30. Secondary Outcome: C24 of ABC in Plasma in Part 1
Description: as for outcome 4
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per millilter | 4.862 (45) | 4.491 (56) | 4.274 (26)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0251, 90% CI 2-sided [0.8480 to 1.2392] — Treatment comparison between Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) and Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, 1 conventional tablet) is presented
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9181, 90% CI 2-sided [0.7592 to 1.1103] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.1165, 90% CI 2-sided [0.9376 to 1.3295] — Treatment comparison between Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) and Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) is presented

31. Secondary Outcome: Ct of ABC in Plasma in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per milliliter | 6.852 (74) | 4.788 (58) | 5.466 (55)

32. Secondary Outcome: T½ of ABC in Plasma in Part 1
Description: as for outcome 25
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 2.314 (30) | 2.525 (26) | 2.382 (29)

33. Secondary Outcome: AUC(0-24) of 3TC in Plasma in Part 1
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of 3TC in Part 1. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours*microgram per milliliter | 11.968 (26) | 11.927 (26) | 10.952 (30)

34. Secondary Outcome: Tmax of 3TC in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 2.50 [1.50 to 5.05] | 2.50 [1.00 to 4.00] | 2.50 [1.50 to 4.08]

35. Secondary Outcome: Tlast of 3TC in Plasma in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 72.00 [48.00 to 72.00] | 72.00 [48.00 to 72.30] | 72.00 [48.00 to 72.02]

36. Secondary Outcome: CL/F of 3TC in Plasma in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters per hour | 22.9237 (26) | 22.9679 (24) | 24.6802 (30)

37. Secondary Outcome: Vz/F of 3TC in Plasma in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Liters | 594.270 (31) | 591.102 (37) | 642.945 (38)

38. Secondary Outcome: C24 of 3TC in Plasma in Part 1
Description: as for outcome 7
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per millilter | 37.963 (29) | 40.913 (24) | 42.434 (27)
Statistical Analysis 1: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets; Test type: Other; Ratio of geometric LS means = 1.0844, 90% CI 2-sided [0.9904 to 1.1873] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.1311, 90% CI 2-sided [1.0334 to 1.2379] — [estimate comment as in outcome 30, analysis 1]
Statistical Analysis 3: Comparison: DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets vs DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 0.9587, 90% CI 2-sided [0.8760 to 1.0493] — [estimate comment as in outcome 1, analysis 3]

39. Secondary Outcome: Ct of 3TC in Plasma in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Nanograms per milliliter | 6.552 (62) | 6.798 (53) | 7.251 (64)

40. Secondary Outcome: T½ of 3TC in Plasma in Part 1
Description: as for outcome 33
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Hours | 17.969 (36) | 17.839 (35) | 18.057 (39)

41. Secondary Outcome: AUC (0-24) of DTG in Plasma in Part 2
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth: Participants received 10 dispersible pediatric DTG/3TC tablets direct-to-mouth
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 35.742 (39) | 61.220 (26) | 46.205 (29)

42. Secondary Outcome: Tmax of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 2.77 [0.50 to 5.00] | 0.77 [0.50 to 4.00] | 1.79 [0.50 to 5.00]

43. Secondary Outcome: Tlast of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 72.00 [48.00 to 72.00] | 72.00 [72.00 to 72.05] | 72.00 [48.00 to 72.05]

44. Secondary Outcome: CL/F of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Liters per hour | 0.9269 (38) | 0.5639 (31) | 0.7300 (32)

45. Secondary Outcome: Vz/F of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Liters | 20.378 (42) | 11.950 (28) | 15.524 (30)

46. Secondary Outcome: C24 of DTG in Plasma in Part 2
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of DTG in Part 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods. Statistics has been presented on geometric LS means.
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Nanograms per millilter | 825.313 (39) | 1289.044 (37) | 1034.078 (33)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 1.5619, 90% CI 2-sided [1.3678 to 1.7835] — Treatment comparison between Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) and Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg, 1 conventional tablet) is presented
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2530, 90% CI 2-sided [1.0973 to 1.4307] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.2466, 90% CI 2-sided [1.0917 to 1.4234] — [estimate comment as in outcome 10, analysis 3]

47. Secondary Outcome: Ct of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Nanograms per milliliter | 95.829 (47) | 131.216 (70) | 107.749 (64)

48. Secondary Outcome: T½ of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 15.238 (21) | 14.690 (18) | 14.741 (23)

49. Secondary Outcome: Tlag of DTG in Plasma in Part 2
Description: as for outcome 41
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 0.00 [0.00 to 0.25] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

50. Secondary Outcome: AUC (0-24) of 3TC in Plasma in Part 2
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters of 3TC in Part 2. Pharmacokinetic analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours*microgram per milliliter | 11.070 (18) | 10.802 (21) | 10.673 (20)

51. Secondary Outcome: Tmax of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 1.00 [0.50 to 3.03] | 1.50 [0.53 to 4.00] | 1.50 [1.00 to 4.00]

52. Secondary Outcome: Tlast of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Hours | 72.00 [72.00 to 72.00] | 72.00 [72.00 to 72.05] | 72.00 [72.00 to 72.05]

53. Secondary Outcome: CL/F of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 18 | 18
Liters per hour | 24.4998 (17) | 24.6933 (21) | 25.1888 (20)

54. Secondary Outcome: Vz/F of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 18 | 18
Liters | 730.859 (17) | 758.790 (28) | 711.280 (22)

55. Secondary Outcome: C24 of 3TC in Plasma in Part 2
Description: as for outcome 13
Time Frame: as for outcome 16
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per millilter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Nanograms per millilter | 35.808 (21) | 38.475 (18) | 38.336 (24)
Statistical Analysis 1: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30 mg Dispersible Tablet; Test type: Other; Ratio of geometric LS means = 1.0745, 90% CI 2-sided [0.9997 to 1.1549] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: DTG 50 mg/3TC 300 mg Tablet vs DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0706, 90% CI 2-sided [0.9961 to 1.1507] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: DTG 5 mg/3TC 30 mg Dispersible Tablet vs DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth; Test type: Other; Ratio of geometric LS means = 1.0036, 90% CI 2-sided [0.9338 to 1.0787] — [estimate comment as in outcome 10, analysis 3]

56. Secondary Outcome: Ct of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Nanograms per milliliter | 7.735 (62) | 8.417 (67) | 7.480 (64)

57. Secondary Outcome: T½ of 3TC in Plasma in Part 2
Description: as for outcome 50
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 18 | 18
Hours | 20.677 (22) | 21.299 (32) | 19.573 (24)

58. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) in Part 1
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. Safety population comprised of all participants enrolled in the study, who took at least one dose of study treatment.
Time Frame: Up to Day 33
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Any AE | 1 | 1 | 2
  Any SAE | 0 | 0 | 0

59. Secondary Outcome: Number of Participants With AEs and Serious Adverse Events SAEs in Part 2
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement.
Time Frame: Up to Day 33
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Any AE | 1 | 0 | 1
  Any SAE | 0 | 0 | 0

60. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 1: Glucose, Calcium, Potassium, Sodium and Urea
Description: Blood samples were collected for the analysis of clinical chemistry parameters which included glucose, calcium, potassium, sodium and urea. All participants population included all participants who received at least one dose of study medication. This population corresponded to all participants enrolled.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Millimoles per liter
  Glucose | 5.031 (0.3501) | 4.931 (0.3448) | 4.933 (0.3709)
  Calcium | 2.377 (0.0577) | 2.371 (0.0775) | 2.384 (0.0704)
  Potassium | 4.31 (0.269) | 4.26 (0.243) | 4.28 (0.271)
  Sodium | 138.1 (2.19) | 138.2 (1.48) | 138.1 (1.55)
  Urea | 4.096 (0.9369) | 4.293 (1.1218) | 4.203 (1.0572)

61. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 1: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotranferase (AST) and Creatinine Phosphokinase (CPK)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CPK.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
International units per Liter
  ALT | 15.3 (7.20) | 14.8 (5.47) | 15.3 (5.80)
  ALP | 54.4 (16.22) | 55.1 (16.89) | 54.4 (16.99)
  AST | 16.1 (3.35) | 16.1 (3.51) | 15.9 (3.29)
  CPK | 90.7 (57.16) | 81.9 (39.34) | 95.8 (52.83)

62. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 1: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including albumin and protein.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Grams per liter
  Albumin | 43.2 (2.82) | 42.9 (2.76) | 43.8 (2.58)
  Protein | 70.7 (4.55) | 70.8 (4.59) | 71.9 (3.73)

63. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 1: Bilirubin, Creatinine and Direct Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Micromoles per liter
  Bilirubin | 9.58 (3.350) | 9.88 (3.612) | 9.99 (4.066)
  Creatinine | 81.47 (14.774) | 82.73 (13.279) | 83.36 (13.647)
  Direct bilirubin | 1.76 (0.469) | 1.88 (0.549) | 1.94 (0.609)

64. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 2: Glucose, Calcium, Potassium, Sodium and Urea
Description: Blood samples were collected for the analysis of clinical chemistry parameters including glucose, calcium, potassium, sodium and urea.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Millimoles per liter
  Glucose | 4.938 (0.2810) | 4.941 (0.3829) | 4.959 (0.3494)
  Calcium | 2.378 (0.0833) | 2.367 (0.1066) | 2.366 (0.1098)
  Potassium | 4.20 (0.252) | 4.10 (0.188) | 4.09 (0.240)
  Sodium | 138.2 (1.50) | 138.3 (1.81) | 138.3 (1.56)
  Urea | 4.603 (0.7878) | 4.343 (0.8311) | 4.398 (0.8430)

65. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 2: ALT, ALP, AST and CPK
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CPK.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
International units per liter
  ALT | 16.1 (11.34) | 15.6 (8.25) | 14.9 (7.44)
  ALP | 60.0 (18.87) | 58.8 (17.53) | 58.9 (17.72)
  AST | 16.5 (5.93) | 15.6 (3.97) | 15.7 (4.96)
  CPK | 90.9 (36.86) | 86.4 (33.82) | 81.7 (25.51)

66. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 2: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including albumin and protein.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Grams per liter
  Albumin | 43.9 (3.02) | 43.1 (4.09) | 43.1 (3.50)
  Protein | 72.1 (3.79) | 70.9 (4.11) | 71.2 (5.26)

67. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters Measured in Part 2: Bilirubin, Creatinine and Direct Bilirubin
Description: as for outcome 63
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Micromoles per liter
  Bilirubin | 10.71 (2.872) | 10.60 (3.275) | 10.58 (2.869)
  Creatinine | 87.66 (16.430) | 87.97 (14.906) | 87.11 (16.453)
  Direct bilirubin | 2.14 (0.451) | 2.11 (0.514) | 2.12 (0.528)

68. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 1: Glucose, Calcium, Potassium, Sodium and Urea
Description: Blood samples were collected for the analysis of clinical chemistry parameters including glucose, calcium, potassium, sodium and urea. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Millimoles per liter
  Glucose | 0.045 (0.4204) | -0.068 (0.3312) | -0.115 (0.3774)
  Calcium | 0.023 (0.0701) | 0.026 (0.0696) | 0.026 (0.0535)
  Potassium | 0.18 (0.256) | 0.17 (0.306) | 0.12 (0.411)
  Sodium | -1.0 (1.73) | -1.0 (1.46) | -0.6 (1.34)
  Urea | 0.361 (0.8156) | 0.386 (0.8436) | 0.027 (1.1490)

69. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 1: ALT, ALP, AST and CPK
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CPK. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
International units per Liter
  ALT | -0.3 (1.69) | -0.1 (2.05) | -0.9 (1.51)
  ALP | -2.6 (6.71) | -0.5 (2.81) | -0.2 (3.84)
  AST | -1.4 (1.62) | -0.6 (1.58) | -1.6 (2.93)
  CPK | -38.2 (65.11) | -25.1 (31.53) | -48.8 (83.77)

70. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 1: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including albumin and protein. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Grams per liter
  Albumin | 0.4 (2.06) | -0.3 (1.61) | 0.4 (1.94)
  Protein | 1.9 (3.31) | 1.6 (3.12) | 2.1 (2.96)

71. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 1: Bilirubin, Creatinine and Direct Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters including bilirubin, creatinine and direct bilirubin. Day -1 was defined as Baseline for clinical chemistry parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Micromoles per liter
  Bilirubin | 1.95 (2.482) | 2.20 (2.313) | 1.63 (2.479)
  Creatinine | 13.61 (5.090) | 13.06 (4.805) | 13.62 (3.782)
  Direct bilirubin | 0.20 (0.409) | 0.30 (0.361) | 0.26 (0.455)

72. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 2: Glucose, Calcium, Potassium, Sodium and Urea
Description: as for outcome 68
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Millimoles per liter
  Glucose | -0.128 (0.3363) | -0.107 (0.3500) | -0.175 (0.4178)
  Calcium | 0.016 (0.0708) | 0.019 (0.0687) | -0.004 (0.0846)
  Potassium | 0.06 (0.268) | -0.02 (0.411) | -0.11 (0.347)
  Sodium | -0.7 (1.93) | -1.3 (1.78) | -0.6 (2.38)
  Urea | 0.176 (1.0267) | 0.084 (1.1918) | 0.414 (0.8744)

73. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 2: ALT, ALP, AST and CPK
Description: as for outcome 69
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
International units per liter
  ALT | -1.2 (3.26) | -2.0 (3.40) | -0.9 (2.85)
  ALP | -1.7 (5.24) | -3.4 (6.06) | -0.7 (4.13)
  AST | -2.1 (3.49) | -2.9 (3.61) | -2.2 (3.73)
  CPK | -34.2 (38.44) | -40.3 (41.91) | -33.2 (30.98)

74. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 2: Albumin and Protein
Description: as for outcome 70
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Grams per liter
  Albumin | -0.1 (2.15) | -0.1 (2.54) | -0.6 (2.45)
  Protein | 1.1 (4.32) | 1.1 (4.30) | 0.6 (4.20)

75. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters Measured in Part 2: Bilirubin, Creatinine and Direct Bilirubin
Description: as for outcome 71
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Micromoles per liter
  Bilirubin | 1.84 (1.974) | 1.56 (2.848) | 1.91 (2.563)
  Creatinine | 10.08 (7.023) | 10.32 (6.185) | 10.83 (6.796)
  Direct bilirubin | 0.22 (0.352) | 0.20 (0.470) | 0.26 (0.434)

76. Secondary Outcome: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelets in Part 1
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelets in Part 1 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
10^9 cells per liter
  Basophils | 0.042 (0.0160) | 0.042 (0.0129) | 0.037 (0.0141)
  Eosinophils | 0.152 (0.1202) | 0.145 (0.0996) | 0.144 (0.1151)
  Lymphocytes | 1.709 (0.4699) | 1.639 (0.4326) | 1.672 (0.5362)
  Monocytes | 0.448 (0.1305) | 0.436 (0.1550) | 0.432 (0.1002)
  Neutrophils | 3.505 (1.2385) | 3.395 (1.5325) | 3.647 (1.2145)
  Leukocytes | 5.86 (1.452) | 5.66 (1.670) | 5.93 (1.410)
  Platelets | 248.8 (64.36) | 247.1 (59.94) | 258.5 (67.34)

77. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Hemoglobin in Part 1
Description: Blood samples were collected for the analysis erythrocyte mean corpuscular hemoglobin in Part 1 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Picograms | 28.11 (2.625) | 27.98 (2.580) | 28.21 (2.585)

78. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Hemoglobin in Part 1
Description: as for outcome 77
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Femtoliter | 83.92 (5.899) | 83.84 (5.810) | 83.97 (5.683)

79. Secondary Outcome: Absolute Values for Erythrocytes in Part 1
Description: Blood samples were collected for the analysis erythrocytes in Part 1 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
10^12 cells per liter | 4.905 (0.4495) | 4.884 (0.4751) | 4.914 (0.4296)

80. Secondary Outcome: Absolute Values for Hemocrit in Part 1
Description: Blood samples were collected for the analysis hemocrit in Part 1 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Percentage of red blood cells in blood | 0.4101 (0.03195) | 0.4076 (0.02824) | 0.4114 (0.03269)

81. Secondary Outcome: Absolute Values for Hemoglobin in Part 1
Description: Blood samples were collected for the analysis hemoglobin in Part 1 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Grams per liter | 137.2 (12.51) | 135.9 (11.13) | 138.1 (13.20)

82. Secondary Outcome: Absolute Values for Hematology Parameters Including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelets in Part 2
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelets in Part 2 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
10^9 cells per liter
  Basophils | 0.042 (0.0186) | 0.044 (0.0253) | 0.039 (0.0171)
  Eosinophils | 0.099 (0.0532) | 0.099 (0.0543) | 0.100 (0.0508)
  Lymphocytes | 1.555 (0.4401) | 1.584 (0.5536) | 1.553 (0.4647)
  Monocytes | 0.373 (0.1229) | 0.378 (0.1367) | 0.369 (0.1264)
  Neutrophils | 2.940 (1.2394) | 2.885 (0.8698) | 2.931 (0.9070)
  Leukocytes | 5.01 (1.513) | 4.98 (1.232) | 4.98 (1.240)
  Platelets | 242.3 (57.86) | 240.6 (58.34) | 244.2 (57.67)

83. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Hemoglobin in Part 2
Description: Blood samples were collected for the analysis erythrocyte mean corpuscular hemoglobin in Part 2 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Picograms | 29.78 (1.582) | 29.79 (1.735) | 29.81 (1.673)

84. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Volume in Part 2
Description: as for outcome 83
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Femtoliter | 88.43 (3.869) | 88.28 (3.867) | 88.34 (4.251)

85. Secondary Outcome: Absolute Values for Erythrocytes in Part 2
Description: Blood samples were collected for the analysis erythrocytes in Part 2 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
10^12 cells per liter | 4.812 (0.4164) | 4.794 (0.4969) | 4.776 (0.4971)

86. Secondary Outcome: Absolute Values for Hemocrit in Part 2
Description: Blood samples were collected for the analysis hemocrit in Part 2 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Percentage of red blood cells in blood | 0.4243 (0.02589) | 0.4219 (0.03425) | 0.4206 (0.03425)

87. Secondary Outcome: Absolute Values for Hemoglobin in Part 2
Description: Blood samples were collected for the analysis hemoglobin in Part 2 at indicated time points.
Time Frame: Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Grams per liter | 143.0 (9.57) | 142.3 (11.33) | 141.8 (11.79)

88. Secondary Outcome: Change From Baseline Values for Hematology Parameters Including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelets in Part 1
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelets in Part 1 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
10^9 cells per liter
  Basophils | -0.009 (0.0176) | -0.009 (0.0162) | -0.011 (0.0100)
  Eosinophils | -0.013 (0.0488) | -0.008 (0.0323) | -0.014 (0.0545)
  Lymphocytes | -0.273 (0.4366) | -0.325 (0.4254) | -0.286 (0.2468)
  Monocytes | -0.082 (0.1001) | -0.066 (0.1332) | -0.098 (0.0818)
  Neutrophils | -0.008 (0.5373) | -0.202 (1.2690) | -0.088 (0.9868)
  Leukocytes | -0.38 (0.640) | -0.61 (1.356) | -0.49 (0.964)
  Platelets | 7.1 (12.27) | -2.8 (13.14) | 3.7 (12.15)

89. Secondary Outcome: Change From Baseline Values for Erythrocyte Mean Corpuscular Hemoglobin in Part 1
Description: Blood samples were collected for the analysis erythrocyte mean corpuscular hemoglobin in Part 1 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Picograms | 0.16 (0.394) | 0.18 (0.303) | 0.19 (0.367)

90. Secondary Outcome: Change From Baseline Values for Erythrocyte Mean Corpuscular Volume in Part 1
Description: as for outcome 89
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Femtoliter | 0.09 (0.756) | 0.09 (0.634) | -0.01 (0.633)

91. Secondary Outcome: Change From Baseline Values for Erythrocytes in Part 1
Description: Blood samples were collected for the analysis erythrocytes in Part 1 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
10^12 cells per liter | 0.191 (0.1562) | 0.121 (0.1513) | 0.221 (0.1443)

92. Secondary Outcome: Change From Baseline Values for Hemocrit in Part 1
Description: Blood samples were collected for the analysis hemocrit in Part 1 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Percentage of red blood cells in blood | 0.0164 (0.01412) | 0.0099 (0.01268) | 0.0188 (0.01373)

93. Secondary Outcome: Change From Baseline Values for Hemoglobin in Part 1
Description: Blood samples were collected for the analysis hemoglobin in Part 1 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Grams per liter | 6.1 (4.19) | 4.0 (4.46) | 7.2 (4.96)

94. Secondary Outcome: Change From Baseline Values for Hematology Parameters Including Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelets in Part 2
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelets in Part 2 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
10^9 cells per liter
  Basophils | -0.004 (0.0134) | -0.004 (0.0142) | -0.008 (0.0142)
  Eosinophils | 0.005 (0.0367) | -0.006 (0.0315) | 0.004 (0.0185)
  Lymphocytes | -0.207 (0.2918) | -0.219 (0.2935) | -0.115 (0.2353)
  Monocytes | -0.074 (0.0668) | -0.079 (0.0608) | -0.049 (0.0972)
  Neutrophils | -0.602 (1.2902) | -0.497 (0.6402) | -0.487 (0.7496)
  Leukocytes | -0.89 (1.333) | -0.81 (0.755) | -0.66 (0.811)
  Platelets | -5.4 (22.31) | 0.3 (14.41) | -2.7 (17.91)

95. Secondary Outcome: Change From Baseline Values for Erythrocyte Mean Corpuscular Hemoglobin in Part 2
Description: Blood samples were collected for the analysis erythrocyte mean corpuscular hemoglobin in Part 2 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Picograms | 0.16 (0.403) | 0.07 (0.353) | -0.04 (0.335)

96. Secondary Outcome: Change From Baseline Values for Erythrocyte Mean Corpuscular Volume in Part 2
Description: as for outcome 95
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Femtoliter | 0.35 (0.678) | -0.01 (0.674) | 0.08 (0.666)

97. Secondary Outcome: Change From Baseline Values for Erythrocytes in Part 2
Description: Blood samples were collected for the analysis erythrocytes in Part 2 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
10^12 cells per liter | 0.201 (0.2539) | 0.224 (0.2171) | 0.179 (0.1813)

98. Secondary Outcome: Change From Baseline Values for Hemocrit in Part 2
Description: Blood samples were collected for the analysis hemocrit in Part 2 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Percentage of red blood cells in blood | 0.0193 (0.02273) | 0.0195 (0.01974) | 0.0159 (0.01427)

99. Secondary Outcome: Change From Baseline Values for Hemoglobin in Part 2
Description: Blood samples were collected for the analysis hemoglobin in Part 2 at indicated time points. Day -1 was defined as Baseline for hematology parameters. Change from Baseline is calculated as the value at specified time point minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Gram per liter | 6.9 (7.70) | 6.8 (5.52) | 5.1 (5.63)

100. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameter in Part 1
Description: The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters can be read as increased, decreased, increase to trace, 1+ and 3+ indicating proportional concentrations in the urine sample. Only participants with abnormal findings for urinalysis at any visit has been presented.
Time Frame: Up to Day 33
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Glucose, No change/decrease | 17 | 17 | 18
  Glucose, Any increase | 0 | 0 | 0
  Ketones, No change/decrease | 17 | 16 | 17
  Ketones, Increase to trace | 0 | 1 | 1
  Occult blood, No change/decrease | 16 | 17 | 16
  Occult blood, Increase to trace | 0 | 0 | 0
  Occult blood, Increase to 1+ | 1 | 0 | 1
  Occult blood, Increase to 3+ | 0 | 0 | 1
  Protein, No change/decrease | 17 | 17 | 18
  Protein, Any increase | 0 | 0 | 0

101. Secondary Outcome: Number of Participants With Urine Potential of Hydrogen (pH)-Part 1
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0).
Time Frame: Up to Day 33
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Participants
  No change/decrease | 14 | 14 | 15
  Any increase | 3 | 3 | 3
  Increase to 5.5 | 1 | 0 | 1
  Increase to 6.0 | 0 | 0 | 0
  Increase to 6.5 | 1 | 1 | 1
  Increase to 7.0 | 1 | 2 | 0
  Increase to 7.5 | 0 | 0 | 0
  Increase to 8.0 | 0 | 0 | 1

102. Secondary Outcome: Number of Participants With Abnormal Urinalysis Parameter in Part 2
Description: as for outcome 100
Time Frame: Up to Day 33
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Glucose, No change/decrease | 18 | 18 | 18
  Glucose, Any increase | 0 | 0 | 0
  Ketones, No change/decrease | 17 | 18 | 18
  Ketones, Increase to trace | 1 | 0 | 0
  Occult blood, No change/decrease | 18 | 17 | 16
  Occult blood Any increase | 0 | 1 | 2
  Occult blood, Increase to trace | 0 | 0 | 1
  Occult blood, Increase to 1+ | 0 | 0 | 0
  Occult blood, Increase to 3+ | 0 | 1 | 1
  Protein, No change/decrease | 18 | 18 | 18
  Protein, Any increase | 0 | 0 | 0

103. Secondary Outcome: Number of Participants With Urine Potential of Hydrogen (pH)-Part 2
Description: as for outcome 101
Time Frame: Up to Day 33
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Participants
  No change/decrease | 11 | 16 | 13
  Any increase | 7 | 2 | 5
  Increase to 5.5 | 0 | 0 | 0
  Increase to 6.0 | 1 | 0 | 1
  Increase to 6.5 | 0 | 0 | 2
  Increase to 7.0 | 4 | 2 | 2
  Increase to 7.5 | 2 | 0 | 0
  Increase to 8.0 | 0 | 0 | 0

104. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings in Part 1
Description: Full 12-lead ECGs were recorded with the participant in a supine position. Absolute QTc Interval: >450, absolute PR Interval: <110 and Absolute QRS Interval: <75 were considered to be potential clinically significant ECG finding. The number of participants with abnormal clinically significant ECG findings are presented.
Time Frame: Baseline (Day -1)
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Participants
  Not clinically significant | 1 | 0 | 1
  Clinically significant | 0 | 0 | 0

105. Secondary Outcome: Number of Participants With Abnormal ECG Findings in Part 2
Description: as for outcome 104
Time Frame: Baseline (Day -1)
Population: All Participants Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Participants
  Not clinically significant | 1 | 1 | 2
  Clinically significant | 0 | 0 | 0

106. Secondary Outcome: Absolute Values for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) of Part 1
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Millimeters of mercury
  SBP, Day 1- 4hours | 117.5 (12.25) | 120.7 (15.73) | 118.9 (10.05)
  SBP, Day 2 | 114.0 (9.50) | 115.2 (11.27) | 115.7 (9.09)
  DBP, Day 1- 4hours | 70.9 (10.88) | 74.0 (11.77) | 71.6 (8.71)
  DBP, Day 2 | 68.1 (8.55) | 68.2 (7.49) | 68.3 (8.20)

107. Secondary Outcome: Absolute Values for Pulse Rate in Part 1
Description: Pulse rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Beats per minute
  Day 1- 4hours | 59.5 (8.32) | 61.6 (12.02) | 59.7 (9.29)
  Day 2 | 63.5 (8.21) | 66.6 (10.04) | 67.4 (9.60)

108. Secondary Outcome: Absolute Values for Temperature in Part 1
Description: Temperature of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention dose and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Degree celsius
  Day 1- 4hours | 36.46 (0.433) | 36.44 (0.411) | 36.51 (0.362)
  Day 2 | 36.41 (0.372) | 36.71 (0.347) | 36.66 (0.415)

109. Secondary Outcome: Absolute Values for SBP and DBP of Part 2
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention dose and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Millimeters of mercury
  SBP, Day 1- 4hours | 116.2 (7.38) | 118.9 (13.31) | 119.1 (13.73)
  SBP, Day 2 | 116.0 (8.01) | 115.5 (9.20) | 113.2 (11.62)
  DBP, Day 1-4 hours | 70.1 (9.38) | 70.9 (11.59) | 71.7 (11.02)
  DBP, Day 2 | 69.5 (6.49) | 71.1 (9.62) | 69.9 (11.46)

110. Secondary Outcome: Absolute Values for Pulse Rate in Part 2
Description: Pulse rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention dose and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Beats per minute
  Day 1-4hours | 63.9 (14.95) | 62.6 (11.25) | 63.3 (13.64)
  Day 2 | 67.7 (14.56) | 64.9 (12.36) | 66.5 (11.42)

111. Secondary Outcome: Absolute Values for Temperature in Part 2
Description: Temperature of participants were measured at indicated time points in semi-supine position after 5 minutes rest.
Time Frame: Day 1 at 4 hours post intervention dose and Day 2 of each treatment period
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Degree celsius
  Day 1-4hours | 36.31 (0.381) | 36.28 (0.373) | 36.39 (0.429)
  Day 2 | 36.33 (0.401) | 36.35 (0.228) | 36.45 (0.343)

112. Secondary Outcome: Change From Baseline in SBP and DBP of Part 1
Description: Blood pressure of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Millimeters of mercury
  SBP, Day 1- 4hours | 0.1 (9.90) | 3.9 (10.59) | 3.1 (8.54)
  SBP, Day 2 | -3.4 (5.94) | -1.6 (7.33) | -0.2 (7.74)
  DBP, Day 1- 4hours | -3.2 (9.36) | 4.6 (8.08) | 1.3 (6.51)
  DBP, Day 2 | -6.1 (5.21) | -1.2 (5.23) | -1.9 (4.89)

113. Secondary Outcome: Change From Baseline in Pulse Rate of Part 1
Description: Pulse rate of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Beats per minute
  Day 1- 4hours | -5.5 (7.31) | -4.4 (5.91) | -7.8 (8.47)
  Day 2 | -1.5 (5.97) | 0.5 (7.37) | -0.1 (8.79)

114. Secondary Outcome: Change From Baseline in Temperature of Part 1
Description: Temperature of participants were measured at indicated time points in semi-supine position after 5 minutes rest. Day 1 (Pre-dose) value was defined as Baseline for vital sign parameters. Change from Baseline value is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets | DTG 5 mg/ABC 60 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 17 | 17 | 18
Degree celsius
  Day 1- 4hours | 0.14 (0.550) | 0.02 (0.256) | 0.21 (0.454)
  Day 2 | 0.09 (0.365) | 0.28 (0.251) | 0.36 (0.412)

115. Secondary Outcome: Change From Baseline in SBP and DBP of Part 2
Description: as for outcome 112
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Millimeters of mercury
  SBP, Day 1- 4hours | -4.4 (7.66) | 0.9 (14.51) | -2.4 (8.63)
  SBP, Day 2 | -4.6 (11.43) | -2.5 (11.95) | -8.3 (9.86)
  DBP, Day 1-4 hours | -0.9 (5.79) | 0.5 (7.73) | -0.5 (7.82)
  DBP, Day 2 | -1.5 (6.69) | 0.7 (6.86) | -2.2 (7.77)

116. Secondary Outcome: Change From Baseline in Pulse Rate in Part 2
Description: as for outcome 113
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Beats per minute
  Day 1-4hours | -4.7 (7.54) | -5.7 (9.38) | -8.6 (13.61)
  Day 2 | -0.9 (7.76) | -3.3 (9.98) | -5.4 (14.18)

117. Secondary Outcome: Change From Baseline in Temperature in Part 2
Description: as for outcome 114
Time Frame: Baseline (Day 1, pre-dose), Day 1- 4 hours and Day 2
Population: All Participants Population.
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | DTG 50 mg/3TC 300 mg Tablet | DTG 5 mg/3TC 30 mg Dispersible Tablet | DTG 5 mg/3TC 30mg Dispersible Tablet Direct to Mouth
Number analyzed (Participants) | 18 | 18 | 18
Degree celsius
  Day 1-4hours | -0.01 (0.508) | 0.05 (0.660) | -0.02 (0.514)
  Day 2 | 0.02 (0.522) | 0.12 (0.565) | 0.03 (0.469)

ADVERSE EVENTS:
Time Frame: The SAEs and AEs were collected from Day 1 up to Day 33.
Description: AEs and SAEs were collected in the Safety Population.
Groups:
- DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet-Part 1: Participants received adult TRIUMEQ as 1 conventional tablet administered as direct-to-mouth.
- DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets-Part 1: Participants received pediatric TRIUMEQ as 10 dispersible tablets administered as dispersion and taken immediately.
- DTG5mg/ABC60mg/3TC30mgdispersible Tablet Direct to Mouth-Part1: Participants received pediatric TRIUMEQ as 10 dispersible tablets administered as direct-to-mouth.
- DTG 50 mg/3TC 300 mg Tablet-Part 2: Participants received adult DTG and 3TC as one conventional tablet direct-to-mouth
- DTG 5 mg/3TC 30 mg Dispersible Tablet-Part 2: Participants received 10 dispersible pediatric DTG/3TC tablets as dispersion
- DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth-Part 2: Participants received 10 dispersible pediatric DTG/3TC tablets direct-to-mouth
Arm/Group | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet-Part 1 | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets-Part 1 | DTG5mg/ABC60mg/3TC30mgdispersible Tablet Direct to Mouth-Part1 | DTG 50 mg/3TC 300 mg Tablet-Part 2 | DTG 5 mg/3TC 30 mg Dispersible Tablet-Part 2 | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth-Part 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/17 | 1/17 | 2/18 | 1/18 | 0/18 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 50 mg/ABC 600 mg/3TC 300 mg Tablet-Part 1 (N=17) | DTG 5 mg/ABC 60 mg/3TC 30 mg Dispersible Tablets-Part 1 (N=17) | DTG5mg/ABC60mg/3TC30mgdispersible Tablet Direct to Mouth-Part1 (N=18) | DTG 50 mg/3TC 300 mg Tablet-Part 2 (N=18) | DTG 5 mg/3TC 30 mg Dispersible Tablet-Part 2 (N=18) | DTG 5 mg/3TC 30 mg Dispersible Tablet Direct to Mouth-Part 2 (N=18)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03441984/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03441984/SAP_001.pdf